CLINICAL TRIAL: NCT06098976
Title: Dental Plaque Removal Around Orthodontic Braces in Adolescents by Water Jet Device Versus Manual Toothbrush: A Randomized Controlled Trial
Brief Title: The Effectiveness of the Water Jet Device in Removing Dental Plaque Around Orthodontic Braces in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UDDS-Pedo-02-2023
Record Dates: First submitted 2023-03-20; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Plaque, Dental
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Jet (Experimental): The patients were taught how to clean their teeth with the Water Jet device (Water Jet, JollyDent, Damascus, Syria) before starting the dental cleaning procedures. Special heads for patients undergoing orthodontic treatment provided by the company were used with each device. The patient applied the Water Jet device on each tooth separately for 10 seconds starting from the upper jaw to the lower jaw.
  Interventions: Device: Water Jet
- Manual toothbrush (Active Comparator): Manual toothbrush: The patients were taught to use the modified vertical method, and the patient brushed the teeth of the upper and lower jaws using traditional toothbrushes (Diamond, JolleyDent, Damascus, Syria), and anti-plaque toothpaste (Elgydium, UniPharma Co., Ltd, Ashrafiyat Sahnaya, Syria).
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Water Jet — The water jet works by directing a stream of water towards the gap between your teeth. The stream of water helps to loosen and remove plaque and food particles stuck in this area.
  Arms: Water Jet
Device: Manual toothbrush — Manual toothbrush: The patients were taught to use the modified vertical method, and the patient brushed the teeth of the upper and lower jaws using traditional toothbrushes (Diamond, JolleyDent, Damascus, Syria), and anti-plaque toothpaste (Elgydium, UniPharma Co., Ltd, Ashrafiyat Sahnaya, Syria).
  Arms: Manual toothbrush

SUMMARY:
The aim of this study was to evaluate the effectiveness of the water jet in removing dental plaque around the orthodontic braces in adolescents.

DETAILED DESCRIPTION:
The aim of this randomized controlled trial was to evaluate the effectiveness of the water jet in removing dental plaque around the orthodontic braces compared to manual toothbrush in adolescents. The null hypothesis was that no significant difference would be noted between the Water Jet and manual toothbrush in removing dental plaque around the orthodontic braces. Such studies provide another dental care tools for maintaining oral hygiene among orthodontic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children.
2. Children aged 11 to 15 years.
3. Children who did not receive any fluoride treatment in the dental clinic.
4. Patients who had orthodontic braces at least on the anterior segment of the upper and lower jaws.

Exclusion Criteria:

1. Special Health Care Needs (SHCN) patients.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Change in Orthodontic Plaque Index | First assessment time: one day before the commencement of the trial. Second assessment time: four months after the commencement of orthodontic treatment
  The plaque accumulation is measured using the Orthodontic Plaque Index (OPI) Dental plaque is going to be disclosed using a disclosing solution (Mira-2-Ton®, Hager & Werken GmbH & Co. KG, Duisburg, Germany) after the last brushing then immediately after cleansing.
  The dentition is divided into sextants, and the highest score of plaque accumulation per sextant is going to be assigned. The OPI for a patient was determined by calculating the average.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Bshara, DDS MSc PhD, Study Chair — gmmn2012@gmail.com
Locations (1):
- Faculty of Dentistry, Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun F, Ahmed A, Wang L, Dong M, Niu W. Comparison of oral microbiota in orthodontic patients and healthy individuals. Microb Pathog. 2018 Oct;123:473-477. doi: 10.1016/j.micpath.2018.08.011. Epub 2018 Aug 8. PMID 30096429
- [Background] Hohoff A, Stamm T, Kuhne N, Wiechmann D, Haufe S, Lippold C, Ehmer U. Effects of a mechanical interdental cleaning device on oral hygiene in patients with lingual brackets. Angle Orthod. 2003 Oct;73(5):579-87. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 14580027
- [Background] Mazzoleni S, De Stefani A, Bordin C, Balasso P, Bruno G, Gracco A. Dental water jet efficacy in the plaque control of orthodontic patients wearing fixed appliance: A randomized controlled trial. J Clin Exp Dent. 2019 Nov 1;11(11):e957-e963. doi: 10.4317/jced.55411. eCollection 2019 Nov. PMID 31700567
- [Background] Ko-Adams C, Cioffi I, Dufour D, Nainar SMH, Levesque CM, Gong SG. Short-term effects of fixed orthodontic appliance on concentrations of mutans streptococci and persister cells in adolescents. Am J Orthod Dentofacial Orthop. 2020 Mar;157(3):385-391. doi: 10.1016/j.ajodo.2019.04.033. PMID 32115117
- [Result] Lopatiene K, Borisovaite M, Lapenaite E. Prevention and Treatment of White Spot Lesions During and After Treatment with Fixed Orthodontic Appliances: a Systematic Literature Review. J Oral Maxillofac Res. 2016 Jun 30;7(2):e1. doi: 10.5037/jomr.2016.7201. eCollection 2016 Apr-Jun. PMID 27489605